CLINICAL TRIAL: NCT04860596
Title: The Effectiveness of Collaborative Health Management Model on Heart Failure Patient Functional Status, Quality of Life, and Rehospitalization: Randomized Controlled Trial
Brief Title: The Effectiveness of Collaborative Health Management Model on Heart Failure Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Antai Medical Care Corperation Antai Tian-Sheng Memorial Hospital/ Department of Nursing/National Ta (Other)
Responsible Party: Principal Investigator, Chih-Wen Chen, Nurse Practitioner Leader, Antai Medical Care Corperation Antai Tian-Sheng Memorial Hospital/ Department of Nursing/National Ta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TSMH IRB No 20-128-B
Record Dates: First submitted 2021-04-18; First posted 2021-04-27 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- collaborative health management model program (Experimental): nursing education and self care program
  Interventions: Behavioral: collaborative health management model
- Routine care (No Intervention): Tranditional education program

INTERVENTIONS:
Behavioral: collaborative health management model — nursing education program
  Arms: collaborative health management model program

SUMMARY:
The purpose of this study is to explore the effect of the collaborative health management model on the functional status, quality of life and rehospitalization rate of patients with heart failure. This is a three-year project. The first phase (introduction phase): A systematic literature review and meta-analysis of collaborative care and heart failure patients will be conducted, and relevant research results will be evaluated for the clinical benefits of heart failure patients, and empirical knowledge will be proposed as The basic holistic conclusions are supported by the research literature on the establishment of a collaborative health management model for heart failure (CHMM). The second stage (construction period): based on the results of systematic literature review and meta-analysis, adopt the CHMM model, design intervention measures, and conduct pilot studies to determine the safety and feasibility of the research, and review future research improvements Wherever possible, develop more complete intervention measures. The third stage (operation period): Randomized controlled trials were adopted, with random sampling and double-blind research design. In the cardiology ward of a regional teaching hospital in the south, 120 patients with heart failure who met the admission criteria were selected, and 60 patients were selected as control group. The group received routine care in the hospital, and 60 of the experimental group received interventions in the collaborative health management model. Data collection includes variables such as physiological indices, functional status, self-care behavior, quality of life, re-admission rate, medical cost. Instruments tools include Minnesota Heart Failure Quality of Life Questionnaire, European Heart Failure Self-care Behavior Scale after the intervention 1 month, 2 months, and 3 months.The intervention effect will be statistically verified and analyzed by GEE. It is hoped that this care model will be applied to the clinical care of patients with heart failure, and will be verified by clinical benefits, reduce symptom troubles, improve quality of life, and reduce medical costs.

DETAILED DESCRIPTION:
The purpose of this study is to explore the effect of the collaborative health management model on the functional status, self care, depression, quality of life and rehospitalization rate of patients with heart failure. This is a three-year project. The first phase (introduction phase): A systematic literature review and meta-analysis of collaborative care and heart failure patients will be conducted, and relevant research results will be evaluated for the clinical benefits of heart failure patients, and empirical knowledge will be proposed as The basic holistic conclusions are supported by the research literature on the establishment of a collaborative health management model for heart failure (CHMM). The second stage (construction period): based on the results of systematic literature review and meta-analysis, adopt the CHMM model, design intervention measures, and conduct pilot studies to determine the safety and feasibility of the research, and review future research improvements Wherever possible, develop more complete intervention measures. The third stage (operation period): Randomized controlled trials were adopted, with random sampling and double-blind research design. In the cardiology ward of a regional teaching hospital in the south, 120 patients with heart failure who met the admission criteria were selected, and 60 patients were selected as control group. The group received routine care in the hospital, and 60 of the experimental group received interventions in the collaborative health management model, including identifying high-risk patients and tracking them by electronic medical records, inter-disciplinary team members discussing patient issues, setting goals together, and passing cross-team members Jointly provide professional care, post-discharge outpatient and telephone follow-up case self-monitoring status, provide telephone consultation hotline, Data collection includes variables such as functional status, self-care behavior, depression, quality of life, re-admission rate. Instruments tools include European Heart Failure Self-care Behavior Scale, Beck Depression Inventory, Minnesota Heart Failure Quality of Life Questionnaire, after the intervention 1 month, 2 months, and 3 months.The intervention effect will be statistically verified and analyzed by GEE. It is hoped that this care model will be applied to the clinical care of patients with heart failure, and will be verified by clinical benefits, reduce symptom troubles, improve quality of life, and reduce medical costs.

ELIGIBILITY:
Inclusion Criteria:

* ⑴Patients diagnosed as heart failure by specialists (NYHA Ⅰ-III); ⑵20 years of age or older; ⑶Patients with clear consciousness and no cognitive impairment and major diseases (such as cancer); ⑷Can communicate in Mandarin and Taiwanese; ⑸ Those who can answer the questionnaire by themselves or with the assistance of a research assistant.

Exclusion Criteria:

* NIL

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
CHF functional status | pre intervenation
  NYHAClass Ⅰ~Ⅲ
CHF functional status | post intervention 1 months
  NYHAClass Ⅰ~Ⅲ
CHF functional status | post intervention 2 months
  NYHAClass Ⅰ~Ⅲ
CHF functional status | post intervention 3 months
  NYHAClass Ⅰ~Ⅲ
CHF quality of life | pre intervention
  Minnesota living with heart failure questionnaire, MLHFQ
CHF quality of life | post intervention 1 months
  Minnesota living with heart failure questionnaire, MLHFQ
CHF quality of life | post intervention 2 months
  Minnesota living with heart failure questionnaire, MLHFQ
CHF quality of life | post intervention 3 months
  Minnesota living with heart failure questionnaire, MLHFQ
CHF rehospitalization | pre intervention
  Re-admission rate
CHF rehospitalization | post intervention 1 months
  Re-admission rate
CHF rehospitalization | post intervention 2 months
  Re-admission rate
CHF rehospitalization | post intervention 3 months
  Re-admission rate
CHF Self care behaviour | pre intervention
  Heart Failure Self-Care Behaviour Sacle, EHFScBS
CHF Self care behaviour | post intervention 1 months
  Heart Failure Self-Care Behaviour Sacle, EHFScBS
CHF Self care behaviour | post intervention 2 months
  Heart Failure Self-Care Behaviour Sacle, EHFScBS
CHF Self care behaviour | post intervention 3 months
  Heart Failure Self-Care Behaviour Sacle, EHFScBS
CHF Depression | pre intervention
  Beck Depression Inventory(BDI)
CHF Depression | post intervention 1 months
  Beck Depression Inventory(BDI)
CHF Depression | post intervention 2 months
  Beck Depression Inventory(BDI)
CHF Depression | post intervention 3 months
  Beck Depression Inventory(BDI)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Wen Chen, Study Chair — employer
Locations (2):
- Taiwan (2):
  - Antai Medical Care Cooperation Antai Tian-Sheng Memorial Hospital, Pingtung City, Donggang Township
  - Research team, Pingtung City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen CW, Wang TJ, Liu CY, Chuang YH, Su CC, Wu SV. Effectiveness of a nurse practitioner-led collaborative health care model on self-care, functional status, rehospitalization and medical costs in heart failure patients: A randomized controlled trial. Int J Nurs Stud. 2025 Feb;162:104980. doi: 10.1016/j.ijnurstu.2024.104980. Epub 2024 Dec 19. PMID 39709786